CLINICAL TRIAL: NCT05607498
Title: A First-in-human, Phase I, Open-Label Study of EMB-07, a Bi-specific Antibody Anti-CD3 and Receptor Tyrosine Kinase-like Orphan Receptor 1 (ROR1) in Patients With Locally Advanced/Metastatic Solid Tumors or Relapse/Refractory Lymphoma
Brief Title: First in Human Study of EMB-07 in Locally Advanced/Metastatic Solid Tumors or Relapse/Refractory Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EpimAb Biotherapeutics (Suzhou)Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMB07X101
Record Dates: First submitted 2022-10-27; First posted 2022-11-07 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-09

CONDITIONS: Advanced/Metastatic Solid Tumors; Relapse/Refractory Lymphoma
Keywords: Phase I; Bispecific antibody; CD3; ROR1; EMB07; Dose escalation; Advanced/Metastatic Solid Tumors; Relapse/Refractory Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMB-07-Patients with solid tumor (Experimental): Patients with solid tumor will receive intravenous infusions of EMB-07 weekly (QW). Dose escalation will continue until the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) is reached or all planned doses are administered.
  Interventions: Drug: EMB07
- EMB07-Patients with lymphoma (Experimental): Patients with lymphoma will receive intravenous infusions of EMB-07 weekly (QW). Dose escalation will continue until the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) is reached or all planned doses are administered.
  Interventions: Drug: EMB07

INTERVENTIONS:
Drug: EMB07 — EMB07 is a MAT-Fab bispecific antibody against CD3 and RORI

SUMMARY:
For solid tumors and lymphoma, respectively: This study is to evaluate the safety and tolerability of EMB-07 and to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D). Pharmacokinetics (PK), immunogenicity, and the anti-multiple myeloma activity of EMB-07 will also be assessed.

DETAILED DESCRIPTION:
This is a phase I, multicenter, open label, dose escalation, first in human study, designed to assess safety and tolerability, and to identify the maximum tolerated dose (MTD) and/or recommended Phase 2 dose for EMB-07 in patient with locally advanced/metastatic solid tumors or relapse/refractory Lymphoma . Pharmacokinetics, pharmacodynamics, immunogenicity and response will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
2. Male or female, and aged ≥ 18 years
3. Treatment group A: Patients with histologically or cytologically locally advanced unresectable or metastatic solid tumors limiting to triple-negative breast cancer, lung adenocarcinoma, ovarian cancer, pancreatic cancer, colorectal cancer, gastric cancer, prostate cancer, bladder cancer, and uterus cancer. Treatment group B: Patients with histologically or cytologically relapse/refractory lymphoma limiting to chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), mantle cell lymphoma (MCL) and diffuse large B cell lymphoma (DLBCL).
4. Treatment group A: Standard therapies do not exist, or are no longer effective, or are not tolerable or accessible to the patient measurable or evaluable disease per RECIST V1.1. Treatment group B: Presence of at least one two-dimensional measurable lesion confirmed by imaging (CT or MRI) (either lymph nodes lesions with any long diameter > 1.5 cm or extranodal lesions with any long diameter > 1.0 cm); for CLL patients whose baseline imaging evaluation determined that no two-dimensional measurable lesions, their peripheral blood monoclonal B lymphocytes should be ≥ 5.0×109/L.
5. Patients must provide archival tumor samples, or a biopsy will be required if archival tumor sample is not available. Archival tumor sample must be taken ≤ 2 years prior to screening, otherwise a fresh tumor biopsy at screening is required.
6. ECOG performance status 0 or 1
7. Adequate organ function to participate in the trial.
8. Recovery from adverse events (AEs) related to prior anticancer therapy.

Exclusion Criteria:

1. Prior treatment with any agent targeting ROR1.
2. History of Grade 4 immune-related adverse events (irAEs) or irAEs requiring discontinuation of prior therapies.
3. Patient with primary central nervous system (CNS) malignancy or symptomatic CNS metastases. Patients with solid tumors with CNS metastases are eligible if they do not need to receive local radiation treatment at the discretion of investigator or if radiation therapy for CNS metastases is completed ≥ 4 weeks prior to study treatment.
4. Anticancer therapy or radiation < 5 half-lives or 4 weeks (whichever is shorter) prior to study treatment.
5. Abuse on alcohol, cannabis-derived products, or other drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events as assessed by CTCAE V5.0. | Screening up to 30 days after the last dose.
  Incidence and severity of AE.
Incidence of serious adverse events (SAE). | Screening up to 30 days after the last dose, or beyond 30 days if SAE is confirmed to be treatment related.
  Incidence of SAE.
Incidence of dose interruptions. | Screening up to 30 days after the last dose.
  Incidence of dose interruptions of EMB-07 during treatment as a measure of tolerability.
Dose intensity. | Screening up to 30 days after the last dose.
  Actual amount of drug taken by patients divided by the planned amount.
The incidence of DLTs during the first cycle of treatment. | First infusion to the end of cycle 1. (each cycle is 28 days).
  The dose limiting toxicities are based on drug related adverse events and are specifically defined in study protocol.

SECONDARY OUTCOMES:
Overall response rate. | From the date of dosing untill the date of first documented progression or date of death from any casue, whichever case first, expected average 6 months.
  Overall response rate measured by RECIST V1.1, iWCLL-2018, Lugano 2014
Area under the serum concentration-time curve (AUC) of EMB-07. | Through treatment until EOT visit, expected average 6 months.
  Blood samples for serum PK analysis will be obtained (AUC).
Maximum serum concentration (Cmax) of EMB-07. | Through treatment until EOT visit, expected average 6 months.
  Blood samples for serum PK analysis will be obtained (Cmax).
Trough concentration (Ctrough) of EMB-07. | Through treatment until EOT visit, expected average 6 months.
  Blood samples for serum PK analysis will be obtained (Ctrough).
Average concentration over a dosing interval (Css, avg) of EMB-07. | Through treatment until EOT visit, expected average 6 months.
  Blood samples for serum PK analysis will be obtained (Css,avg).
Terminal half-life (T1/2) of EMB-07. | Through treatment until EOT visit, expected average 6 months.
  Blood samples for serum PK analysis will be obtained (T1/2).
Systemic clearance (CL) of EMB-07. | Through treatment until EOT visit, expected average 6 months.
  Blood samples for serum PK analysis will be obtained (CL).
Steady state volume of distribution (Vss) of EMB-07. | Through treatment until EOT visit, expected average 6 months.
  Blood samples for serum PK analysis will be obtained (Vss).
Progression free survival (PFS) of EMB-07 as assessed by RECIST 1.1, iWCLL-2018, Lugano 2014 | Through treatment discontinuation: an average of 6 months
  From the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, expected average 6 months.
Incidence and titer of anti-drug antibodies stimulated by EMB-07. | Up to End of Treatment Follow Up Period (30 days after the last dose)
  Antibodies to EMB-07 will be assessed to evaluate potential immunogenicity.

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (2):
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - One Clinical Research, Nedlands, Western Australia
- China (8):
  - Hunan Cancer Hospital, Changsha, Hunan
  - Affiliated Hospital of Hebei University, Baoding
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - The Affiliated Tumour Hospital of Harbin Medical University, Harbin
  - Shandong Cancer Hospital, Shandong
  - Tianjin Medical University Cancer Institue & Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No